CLINICAL TRIAL: NCT05128331
Title: The Effect of sPERMIdine supplemenTation on the Metabolic, Neuronal and Cardiovascular Response to Exercise TRAINING in Patients With Heart Failure With Preserved Ejection Fraction
Brief Title: sPERMIdine supplemenTation on Metabolic, Neuronal and Cardiovascular Response to Exercise TRAINING
Acronym: PERMIT_EX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PERMIT-HGW-DZHK40
Record Dates: First submitted 2021-09-16; First posted 2021-11-22 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2021-09

CONDITIONS: Heart Failure, Diastolic
Keywords: Exercise; Spermidine
MeSH Terms: conditions — Heart Failure, Diastolic; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spermidine supplementation (Experimental): Study participants are provided with spermidine supplementation
  Interventions: Dietary Supplement: spermidineLife
- Placebo supplementation (Placebo Comparator): Study participants are provided with a placebo supplementation
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: spermidineLife — dietary supplement that is made of natural wheat germ extract with high spermidine content
  Arms: Spermidine supplementation
Dietary Supplement: Placebo — dietary supplement that is made of cellulose.
  Arms: Placebo supplementation

SUMMARY:
This study explores whether spermidine supplementation improves the metabolic, neurological-cognitive and cardiovascular response to structured exercise training in patients with heart failure with preserved ejection fraction. The investigators aim to show that a faster adaptation to exercise may improve long term adherence to a more active lifestyle.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction is the largest unmet need in medicine. Exercise training is a pivotal lifestyle intervention which has been shown to have beneficial effects with regards to metabolic, neurological-cognitive and cardiovascular outcomes in these patients. Yet, not every patients responds equally fast to an exercise training intervention. This trial explores whether the supplementation of spermidine can increase the response to a structured aerobic exercise training. The investigators will recruit 30 patients who will either receive a spermidine supplement or a placebo. The study participants are invited for a first follow-up visit after four weeks. The exercise intervention starts at week 5 and continues for 12 weeks. Hence, overall there are three visits (baseline, week four and week twelve).

ELIGIBILITY:
Inclusion Criteria:

* diastolic heart failure (E/e' > 8, left ventricular ejection fraction (LVEF) => 50 %, dyspnea)

Exclusion Criteria:

* nutritional supplements with polyamines
* acute myo-, endo- or pericarditis
* aortic valve stenosis (2nd degree)
* cardiomyopathy or severe left ventricular hypertrophy (Interventricular septal end diastolic thickness or posterior wall thickness > 17 mm)
* AV block (second degree)
* pulmonary hypertension
* thromboembolic event in the last six months
* anemia
* infection (with fever) within the last four weeks
* cancer

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory exercise capacity | 16 weeks
  Change in cardiorespiratory exercise capacity (VO2peak) in ml/min/kg before and after of exercise training

SECONDARY OUTCOMES:
Diastolic function | 16 weeks
  Change in diastolic function based on echocardiography (E/e')
Microvascular function | 16 weeks
  Reactive hyperemia index assessed using EndoPat

OTHER OUTCOMES:
Multiple-Choice Vocabulary Intelligence Test (MWT-B) | 16 weeks
  Multiple-Choice Vocabulary Intelligence Test: Measure: total number of correctly checked lines. Final outcome: IQ (standard value and percentile rank)
Mnemonic Similarity Task (MST) | 16 weeks
  Mnemonic Similarity Task (MST). % of correctly answered tasks (0 - 100 %). final outcome: D - Prime
Verbal Learning and Memory Test (VLMT) | 16 weeks
  Verbal Learning and Memory Test (VLMT) % of correctly answered tasks (0 - 100 %). final outcome: D - Prime
Digit Span test battery for attention testing | 16 weeks
  Digit Span test battery for attention testing; from 0 to 8, Score: maximum number of digits that were correctly remembered after 3 erros the test ends. direction of the task (forward or backwards), the longest sequence successfully reached and passed, and the total number of attempts
brain magnetic resonance imaging (MRI) - T1 | 16 weeks
  brain magnetic resonance imaging (MRI) T1 to assess cortical brain structure pre and post intervention
brain magnetic resonance imaging (MRI) - FLAIR | 16 weeks
  brain magnetic resonance imaging (MRI) - FLAIR to assess white matter hyperintensities pre and post intervention
brain magnetic resonance imaging (MRI) - DTI | 16 weeks
  brain magnetic resonance imaging (MRI) - DTI to assess fractional anisotropy and fiber tracking pre and post intervention
brain magnetic resonance imaging (MRI) - resting state fMRI | 16 weeks
  brain magnetic resonance imaging (MRI) resting state fMRI to assess brain network connectivity pre and post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular examination center of the University Medicine Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No
Our ethics approval does not allow to share IPD for this trial.